CLINICAL TRIAL: NCT04268862
Title: Ethnic Dependence of the Metabolic Defects in Prediabetic Individuals: Kuwaiti Arabs Versus Indians
Brief Title: Metabolic Defects in Prediabetic Kuwaiti Arabs and Indians
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dasman Diabetes Institute (Other)
Responsible Party: Principal Investigator, Dr. Ebaa Al Ozairi, Chief Medical Officer, Dasman Diabetes Institute
Other Study IDs: RA HM-2019-003
Record Dates: First submitted 2019-10-20; First posted 2020-02-13 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Pathophysiology; Metabolic Glucose Disorders
Keywords: Beta cell function; Insulin Resistance; Arabs; Asian Indians
MeSH Terms: conditions — Glucose Metabolism Disorders; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Insulin and C-peptide will be measured in plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Insulin resistance and beta cell dysfunction are the major core defects responsible for the development of type 2 diabetes (T2DM). Although insulin resistance is the early metabolic defect detected in subjects destined to develop T2DM, it is the beta cell failure which is responsible for the development of hyperglycemia.

Longitudinal and cross-sectional studies have demonstrated that, initially, the compensatory hyperinsulinemia is sufficient to offset the insulin resistance and maintain normal glucose tolerance. However, when the beta cell fails to adequately compensate for the insulin resistance, glucose homeostasis deteriorates. Initially, this is manifest as impaired glucose tolerance (IGT) and later as overt diabetes. It follows that the level of beta cell failure at which hyperglycemia becomes evident depends upon the prevailing level of insulin resistance. A more severe insulin resistance results in development of overt hyperglycemia at lower level of beta cell failure. The investigators previously have shown that the severity of insulin resistance varies amongst different ethnic groups (Arabs versus Indians). Thus, the level of beta cell failure at which overt hyperglycemia becomes evident amongst each ethnic group also varies. Thus, individuals/ethnic groups with more severe insulin resistance, overt hyperglycemia becomes evident at lower level of beta cell dysfunction. Conversely, severe beta cell dysfunction is required for evert hyperglycemia to develop in individuals/ethnicities with less severe insulin resistance.

In the present study, the investigators aim to quantitate beta cell function with the gold standard technique (i.e. hyperglycemic clamp) in Arab and Indian non-diabetic individuals and relate the level of beta cell function to the prevailing level of insulin resistance measured as the glucose infusion rate divided by the mean plasma insulin concentration during the clamp.

DETAILED DESCRIPTION:
Insulin resistance and the accompanying hyperinsulinemia also lead to the development of multiple metabolic abnormalities which are responsible, at least in part, for the excessive risk of coronary heart disease in T2DM , non-alcoholic steatohepatitis (NASH), and impaired diastolic left ventricular (LV) function. Thus, insulin resistance contributes, not only to increased T2DM risk, but also to the morbidity and mortality associated with the disease.

Etiology of Insulin Resistance Insulin resistance is closely related to obesity. Multiple mechanisms contribute to insulin resistance in obese individuals. Accumulation of fat in insulin target tissues (i.e. ectopic fat), e.g. in myocytes and hepatocytes, plays a central role in the pathogenesis of insulin resistance. When energy intake exceeds energy expenditure, the energy excess is stored in subcutaneous adipocytes in the form of triglycerides. However, under conditions of persistent positive energy balance, subcutaneous fat stores become filled and the excess energy spills over into the circulation in the form of FFA, leading to increased fat content in lean tissues, i.e. ectopic fat. Many studies have documented the important role of ectopic fat content in the pathogenesis of insulin resistance in obese individuals. The severity of insulin resistance in skeletal muscle and liver strongly correlates with ectopic fat content in myocytes and hepatocytes, respectively. Further, therapies that deplete ectopic fat, e.g. weight loss and pioglitazone, significantly improve insulin sensitivity.

Fat spill over and the subsequent increase in ectopic fat content in lean tissues could result from subcutaneous fat cells that are filled to capacity or the inability of the subcutaneous fat stores to expand. Consistent with this hypothesis, several studies have demonstrated increased fat cell size in subcutaneous fat in insulin resistant obese individuals compared to insulin sensitive controls. Moreover, large fat cells have a higher rate of lipolysis and decreased rate of FFA esterification compared to small fat cells, suggesting decreased ability of large fat cells to further store fat in subcutaneous adipose tissue in obese individuals. Of note, large fat cell size is a strong predictor of future T2DM risk in non-diabetic individuals, independent of insulin resistance. Collectively, these results have led to the hypothesis that inability of subcutaneous fat tissue to expand results in fat spill over into muscle, liver, heart, etc and the subsequent development of insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

1. age 21-65 years
2. BMI=18-45 kg/m2
3. NGT (FPG<100 mg/dl and 2-hour PG <140 mg/dl) or IGT (FPG < 125 mg/dl, and 2-hour PG=140-199 mg/dl) according to the ADA criteria.
4. Good general health as determined by physical exam, medical history, blood chemistries, CBC, TSH, T4, lipid profile.
5. Stable body weight (± 3 lbs) over the preceding three months
6. Not participate in an excessively heavy exercise program.

Exclusion Criteria:

Subjects with

* Haematocrit < 34.0
* Diabetes, Thyroid disorders, Cardiovascular Diseases, Cancer, Bronchial Asthma and any autoimmune disease.
* Subjects who receive medications which affect glucose tolerance, e.g. Steroids
* Subjects who participate in excessively heavy exercise programs, e.g. Athletes

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects from two ethnic groups will participate in the present study: (1) 60 Kuwaiti Arab subjects and (2) 60 subjects of Indian ethnicity. Each ethnic group will include 30 subjects with normal glucose tolerance (NGT), and 30 subjects with impaired glucose tolerance (IGT) according to the American Diabetes Association criteria.
  Subjects in each ethnic group will be matched for age, sex, BMI and family history of type 2 diabetes.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Insulin Resistance | 15 months
  Insulin Resistance measured as total glucose disposal TGD with the Insulin Clamp
Insulin Secretion | 15 months
  First phase and second phase insulin secretion measured with the hyperglycemic clamp
Beta Cell function | 15 months
  Beta cell function for the first phase and second phase measured as ∆C-Pep/(1/TGD)
Comparison of genetic markers | 15 months
  Genetic markers that correlate with the metabolic phenotype measured using GWAS
GLP1 Action | 15 months
  GLP1 Action measured as increase in C-peptide during the hyperglycemic clamp caused by exenatide infusion

CONTACTS AND LOCATIONS:
Overall Officials: Ebaa AlOzairi, MD, PhD, Principal Investigator — Dasman Diabetes Institute
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Kuwait

REFERENCES:
- [Background] Defronzo RA. Banting Lecture. From the triumvirate to the ominous octet: a new paradigm for the treatment of type 2 diabetes mellitus. Diabetes. 2009 Apr;58(4):773-95. doi: 10.2337/db09-9028. No abstract available. PMID 19336687
- [Background] Abdul-Ghani MA, DeFronzo RA. Pathophysiology of prediabetes. Curr Diab Rep. 2009 Jun;9(3):193-9. doi: 10.1007/s11892-009-0032-7. PMID 19490820
- [Background] DeFronzo RA. Insulin resistance, lipotoxicity, type 2 diabetes and atherosclerosis: the missing links. The Claude Bernard Lecture 2009. Diabetologia. 2010 Jul;53(7):1270-87. doi: 10.1007/s00125-010-1684-1. Epub 2010 Apr 2. PMID 20361178
- [Background] Clarke GD, Solis-Herrera C, Molina-Wilkins M, Martinez S, Merovci A, Cersosimo E, Chilton RJ, Iozzo P, Gastaldelli A, Abdul-Ghani M, DeFronzo RA. Pioglitazone Improves Left Ventricular Diastolic Function in Subjects With Diabetes. Diabetes Care. 2017 Nov;40(11):1530-1536. doi: 10.2337/dc17-0078. Epub 2017 Aug 28. PMID 28847910
- [Background] Abdul-Ghani MA, DeFronzo RA. Pathogenesis of insulin resistance in skeletal muscle. J Biomed Biotechnol. 2010;2010:476279. doi: 10.1155/2010/476279. Epub 2010 Apr 26. PMID 20445742
- [Background] Eckel RH, Kahn SE, Ferrannini E, Goldfine AB, Nathan DM, Schwartz MW, Smith RJ, Smith SR. Obesity and type 2 diabetes: what can be unified and what needs to be individualized? J Clin Endocrinol Metab. 2011 Jun;96(6):1654-63. doi: 10.1210/jc.2011-0585. PMID 21602457
- [Background] Lettner A, Roden M. Ectopic fat and insulin resistance. Curr Diab Rep. 2008 Jun;8(3):185-91. doi: 10.1007/s11892-008-0032-z. PMID 18625114
- [Background] Sabag A, Way KL, Keating SE, Sultana RN, O'Connor HT, Baker MK, Chuter VH, George J, Johnson NA. Exercise and ectopic fat in type 2 diabetes: A systematic review and meta-analysis. Diabetes Metab. 2017 Jun;43(3):195-210. doi: 10.1016/j.diabet.2016.12.006. Epub 2017 Feb 2. PMID 28162956
- [Background] Lundgren M, Svensson M, Lindmark S, Renstrom F, Ruge T, Eriksson JW. Fat cell enlargement is an independent marker of insulin resistance and 'hyperleptinaemia'. Diabetologia. 2007 Mar;50(3):625-33. doi: 10.1007/s00125-006-0572-1. Epub 2007 Jan 10. PMID 17216279
- [Background] Weyer C, Foley JE, Bogardus C, Tataranni PA, Pratley RE. Enlarged subcutaneous abdominal adipocyte size, but not obesity itself, predicts type II diabetes independent of insulin resistance. Diabetologia. 2000 Dec;43(12):1498-506. doi: 10.1007/s001250051560. PMID 11151758
- [Background] McLaughlin T, Craig C, Liu LF, Perelman D, Allister C, Spielman D, Cushman SW. Adipose Cell Size and Regional Fat Deposition as Predictors of Metabolic Response to Overfeeding in Insulin-Resistant and Insulin-Sensitive Humans. Diabetes. 2016 May;65(5):1245-54. doi: 10.2337/db15-1213. Epub 2016 Feb 16. PMID 26884438
- [Background] Badoud F, Perreault M, Zulyniak MA, Mutch DM. Molecular insights into the role of white adipose tissue in metabolically unhealthy normal weight and metabolically healthy obese individuals. FASEB J. 2015 Mar;29(3):748-58. doi: 10.1096/fj.14-263913. Epub 2014 Nov 19. PMID 25411437
- [Background] Arner P, Engfeldt P, Ostman J. Relationship between lipolysis, cyclic AMP, and fat-cell size in human adipose tissue during fasting and in diabetes mellitus. Metabolism. 1979 Mar;28(3):198-209. doi: 10.1016/0026-0495(79)90065-9. PMID 216883
- [Background] Scherer PE. The Multifaceted Roles of Adipose Tissue-Therapeutic Targets for Diabetes and Beyond: The 2015 Banting Lecture. Diabetes. 2016 Jun;65(6):1452-61. doi: 10.2337/db16-0339. PMID 27222389
- [Background] Bays H, Mandarino L, DeFronzo RA. Role of the adipocyte, free fatty acids, and ectopic fat in pathogenesis of type 2 diabetes mellitus: peroxisomal proliferator-activated receptor agonists provide a rational therapeutic approach. J Clin Endocrinol Metab. 2004 Feb;89(2):463-78. doi: 10.1210/jc.2003-030723. No abstract available. PMID 14764748